CLINICAL TRIAL: NCT01633905
Title: Electrophysiological Correlates of Emotional and Crossmodal Stimuli Processing Among Alcohol-dependent Participants : Exploration of the Peripheral Presentation Effect
Brief Title: Electrophysiological Correlates of Emotional and Crossmodal Stimuli Processing Among Alcohol-dependent Participants
Acronym: ALCOLAT
Status: Completed | Type: Observational
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Other Study IDs: 2010_01; 2010-A00595-34 (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2011-08-09; First posted 2012-07-04 (Estimated); Last update posted 2015-06-17 (Estimated); Status verified 2015-06

CONDITIONS: Alcohol-dependence
Keywords: alcohol-dependence; event-related potentials; emotion; crossmodal; peripheral processing
MeSH Terms: conditions — Alcoholism

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- alcohol-dependent patients: 22 recently detoxified participants diagnosed as alcohol-dependant on the basis of DSM-IV criteria who will performed an emotion-detection task on unimodal (visual or auditory) or crossmodal (visuo-auditory) stimulations presented centrally or peripherally
- control group: 22 healthy controls without any psychiatric or neurological diagnosis who will performed an emotion-detection task on unimodal (visual or auditory) or crossmodal (visuo-auditory) stimulations presented centrally or peripherally

SUMMARY:
Alcohol-dependence is the most widespread addiction in Western countries and leads to a wide range of impairments at cerebral and cognitive levels. It has also been showed that alcohol-dependence is associated with emotional disturbances, particularly for the decoding of emotional facial expressions (EFE). In view of the crucial role played by EFE to develop and maintain satisfactory interpersonal relations, this emotional processing impairment may have deleterious consequences on alcohol-dependent patient's social well-being, and this deficit is thus of particular clinical interest. Nevertheless, this deficit has up to now been evaluated only by means of experiments using paradigms with low ecological value (i.e. presentation of EFE in isolation and in the central vision field), while in the real life, emotional stimuli are most frequently appearing together with other emotional stimulations (particularly voices) and in the peripheral vision field. Moreover, the cerebral correlates of this emotional deficit are still to be determined.

The present study thus aims at exploring the Emotional Facial Expressions (EFE) decoding in alcoholism using a more ecological paradigm, based on peripheral presentation of emotional crossmodal stimuli (i.e. the simultaneous presentation of emotionally congruent face and voice).

Main aim: Determining the electrophysiological characteristics (latencies and amplitudes) of the event-related components elicited among recently detoxified alcohol-dependent participants, while performing an emotion-detection task on crossmodal stimuli (voices and/or faces) presented centrally or peripherally, and comparing these characteristics with those obtained among paired healthy participants.

Secondary objectives:

* Exploring the electrophysiological pattern modifications among alcohol-dependent participants for the emotional faces and voices decoding (unimodal conditions), using spatio-temporal analyses methods.
* Exploring the electrophysiological waves associated with peripheral crossmodal stimuli processing among healthy participants.
* Exploring the behavioral correlates (reaction times and accuracy) of the emotion-detection task among alcohol-dependent participants while processing peripheral stimuli.
* Exploring the psychopathological comorbidities among alcohol-dependent participants and their influence on the behavioral and electrophysiological results.

DETAILED DESCRIPTION:
Methodology: Evaluation the event-related potentials elicited among alcohol-dependent and healthy participants while performing an emotion-detection task on unimodal (visual or auditory) or crossmodal (visuo-auditory) stimulations presented centrally or peripherally. Event-related potentials allow to monitor the electrical activity of the brain with high temporal resolution and to detect even minor neurocognitive restrictions. This cerebral measures will be completed by behavioral (reaction times and accuracy) and psychopathological measures.

No specific interventions assigned to the subjects of the study.

Evaluations: The room contains a panoramic screen (2.4 X 4 meters) covering a 180 degrees of visual angle. Participants will seat in a chair situated two meters away from the screen, in front of a table on which the response pad will be placed. Three projectors will display the visual stimulations, either centrally or lateralized (-12°, -24°on the left or +12°, +24° on the right). Headphones will be placed on participants' ears in order to display the auditory stimulations, either on both ears or lateralized (left or right ear), and presented separately (unimodal conditions) or simultaneously (crossmodal condition) with the visual stimuli. Visual stimuli, constructed using FaceGen 3.4 program, will be emotional faces (two males, two females) depicting happiness, anger or a neutral expression. Auditory stimuli (two males, two females), from a validated battery, will be emotional voices depicting happiness, anger or a neutral prosody and presented at a 70 decibels level. Crossmodal stimulations will be a combination of visual and auditory stimuli, congruent for gender and emotion. Experiment will be composed of 39 conditions: 3 stimulations (visual, auditory, visuo-auditory) X 3 emotions (anger, happiness, neutral) X 3/5 lateralisation (-24°, -12°, 0°, 12°, 24°). Each condition will be evaluated on the basis of 50 stimulations. Event-related potentials will be recorded during the whole experiment by means of a 128 electrodes cap placed on participant's head and connected with an amplifier (Advanced Neuro Technology, ANT) and a recording computer, synchronised with the stimulation system. Behavioral responses will be recorded by means of a response pad. Psychopathological measures will be conducted using validated questionnaires: State and trait anxiety (STAI A and B, Spielberger et al., 1983), depression (BDI, Beck et al., 1987), interpersonal problems (Horowitz et al. (1988)), evaluating the quantity and quality of the social interactions, and the integration in the family and relationship background and alexithymia (Bagby et al., 1994).

ELIGIBILITY:
Inclusion Criteria :

* for alcohol-dependence group : alcohol-dependent subjects
* for control group : healthy volunteers without psychiatric
* for control group : healthy volunteers without neurological diagnosis

Exclusion Criteria :

* more than 60 years old and less than 18 years old,
* no French-speaking,
* not normal or not corrected-to-normal auditory acuity,
* not normal or not corrected-to-normal visual acuity

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: * 22 recently detoxified participants, diagnosed as alcohol-dependent on the basis of DSM-IV criteria, free of any alcohol consumption during the last 15 days, and without any other DSM-IV criteria
  * 22 healthy controls paired for gender, age and educational level with alcohol-dependent participants, without any alcohol consumption during the last three days and without any psychiatric or neurological diagnosis.
  All participants will be between 18 and 60 years of age, will be French-speaking and will present a normal or corrected-to-normal auditory and visual acuity.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2010-12; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
brain electrical responses amplitudes and latencies | participants will be followed an average of 2 hours for the duration of experiment
  Differences in latencies, mainly the P3b wave, in milliseconds and differences in brain electrical responses amplitudes in millivolts, between the alcohol-dependent group and the healthy participants group.

SECONDARY OUTCOMES:
reactions times | participants will be followed an average of 2 hours for the duration of experiment
  Differences in reactions times during the emotion-detection task between the two groups.
behavioural and psychopathological measures | participants will be followed an average of 2 hours for the duration of experiment
  Differences in anxiety level, psychopathology, interpersonal problems level, alexithymia level, measured by validated questionnaires.
percentage of correct answers | participants will be followed an average of 2 hours for the duration of experiment
  Differences in percentage of correct answers between the two groups.

CONTACTS AND LOCATIONS:
Overall Officials: Olivier COTTENCIN, Principal Investigator — University Hospital, Lille
Locations (1):
- University Hospital, Lille, Lille, France